CLINICAL TRIAL: NCT05236153
Title: Electroanatomic Interactions Between Transcatheter Pulmonary Valve Prostheses and Anatomic Isthmuses in Repaired Tetralogy of Fallot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Edward O'Leary, Staff Physician, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-P00038878
Record Dates: First submitted 2022-01-21; First posted 2022-02-11 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Tetralogy of Fallot; Ventricular Tachycardia; Sudden Cardiac Death
MeSH Terms: conditions — Tetralogy of Fallot; Tachycardia, Ventricular; Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- RV mapping (Other): Participants will undergo a sinus rhythm electroanatomic RV substrate map prior to TPVR.
  Interventions: Diagnostic Test: Electroanatomic substrate mapping

INTERVENTIONS:
Diagnostic Test: Electroanatomic substrate mapping — Participants will undergo a sinus rhythm RV substrate map using the HD Grid catheter (Abbott) and the Ensite X electroanatomic mapping system (Abbott) prior to TPVR.

SUMMARY:
Individuals with repaired Tetralogy of Fallot (rTOF) remain at risk for sudden cardiac death from ventricular tachycardia (VT). Transcatheter pulmonary valve replacement (TPVR) indications continue to broaden, yet its capability to reduce the risk of VT and sudden cardiac death remains unknown. Thus, in a cohort of participants with rTOF who are presenting for TPVR the investigators intend to: (1) quantify and localize right ventricular (RV) isthmuses with abnormal voltage and/or conduction velocity; (2) identify which RV isthmuses are at risk of being "jailed" by TPV prostheses; and (3) explore the feasibility of omnipolar technology to characterize wavefront directionality and differentiate slow conduction from conduction block.

DETAILED DESCRIPTION:
Participants will receive general endotracheal anesthesia or conscious sedation provided by cardiac anesthesiology and usual vascular access as per routine clinical care for TPVR. The TPVR procedure will be performed per routine care independent of study participation or study findings.

Participants who elect to participate in this research study will undergo RV activation and voltage mapping using a diagnostic electrophysiology mapping catheter. Prior to the delivery of the valve prosthesis, a 3-dimensional electroanatomic map (EAM) of the RV with simultaneous omnipolar voltage and activation data in sinus rhythm will be created using a high-density multielectrode mapping catheter (8 Fr Advisor HD Grid, Abbott Cardiovascular) and an EAM system (Ensite X, Abbott Cardiovascular). Pre-procedural CCT or CMR imaging will be overlayed on the EAM using the tricuspid valve annulus, pulmonary valve annulus, and proximal coronary sinus as fiducial markers for registration. The plane of the pulmonary valve annulus and/or the existing pulmonary valve prosthesis will be annotated on the EAM, referencing the merged CCT/CMR and fluoroscopic images. Ventricular pacing at physiologic rates (60-120 bpm) may be performed to assist in differentiating slow conduction from conduction block and confirming areas of scar. No programmed ventricular stimulation pacing with the intention to induce ventricular arrhythmias will be performed. No catheter ablation will be performed.

Following the completion of the study protocol, participants will be followed prospectively for 10 years to evaluate for the development of the following outcomes: documented sustained clinical VT, inducible sustained VT or ventricular fibrillation during intracardiac electrophysiology study, placement of a primary or secondary prevention implantable cardioverter defibrillator (ICD), appropriate ICD shock for VT/VF, and/or sudden cardiac arrest/death. Participant medical records will be reviewed annually for the development of these outcomes. Informed research consent for future medical record review and research team contact with the participant or primary cardiologist will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of tetralogy of Fallot (TOF) or double outlet right ventricle (DORV)
* Referred for transcatheter pulmonary valve replacement (TPVR) per routine clinical indications
* Weight >=25 kg

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-11-03 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Jailed anatomical isthmus area | Immediately after the procedure.
  Percent jailing of each anatomical RV isthmus (jailed area / isthmus area x100)
Future arrhythmic event (composite) | 10 years
  Documented sustained VT, inducible sustained VT/VF at a future EP study, appropriate ICD therapy for VT/VF, sudden cardiac arrest

SECONDARY OUTCOMES:
Presence of any jailed anatomical isthmus | Immediately after the procedure.
  >50% of an anatomical isthmus covered by the TPV prosthesis
Number, location, and dimensions of electroanatomically normal isthmuses. | Immediately after the procedure.
  isthmuses with omnipolar voltage >1.5 mV and conduction velocity >0.5 m/sec
Number, location, and dimensions of electroanatomically abnormal isthmuses. | Immediately after the procedure.
  isthmuses with omnipolar voltage <1.5 mV and conduction velocity <0.5 m/sec

CONTACTS AND LOCATIONS:
Overall Officials: Edward T O'Leary, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided